CLINICAL TRIAL: NCT00230854
Title: An Open Label, Dose Escalation Study of EMZ702 in Combination With Pegylated Interferon and Ribavirin in Patients With Chronic Hepatitis C Genotype 1 Non-responsive to Prior Therapy With Pegylated Interferon and Ribavirin
Brief Title: Study in Non-responder Hepatitis C Genotype 1 Patients With EMZ702, Pegylated Interferon and Ribavirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IET-202
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis C; Hepatitis, Viral, Human
Keywords: hepatitis C; genotype 1; non-responders; viral hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis, Viral, Human; Hepatitis C

INTERVENTIONS:
Drug: EMZ702

SUMMARY:
The purpose of this study is to assess the safety and efficacy of repeated intravenous infusions of EMZ702 in combination with pegylated interferon and ribavirin in patients with chronic hepatitis C genotype 1.

DETAILED DESCRIPTION:
In this study, 28 patients with chronic hepatitis C genotype 1 who have failed previous treatment with pegylated interferon plus ribavirin will be treated. The study treatment will consist of the same type and doses of pegylated interferon and ribavirin to which the patient failed to respond plus EMZ702. EMZ702 will be administered intravenously twice a week during the first 12 weeks of treatment. Thereafter and according to viral response, patients will continue to receive pegylated interferon and ribavirin only for up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) genotype 1
* Previous therapy with pegylated interferon and ribavirin
* Documented previous treatment failure

Exclusion Criteria:

* Hepatic dysfunction
* Coinfection with hepatitis B or HIV
* Other unrelated liver diseases
* Liver cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2005-08; Study Completion 2007-07

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of repeated intravenous infusions of EMZ702 in combination with pegylated interferon and ribavirin in patients with chronic hepatitis C genotype 1

SECONDARY OUTCOMES:
To evaluate the viral response and pharmacokinetic profile of repeated intravenous infusions of EMZ702 in combination with pegylated interferon and ribavirin in patients with chronic hepatitis C genotype 1

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Pastrak, M.D., Study Director — OPKO Health, Inc.
Locations (2):
- Canada (2):
  - L.H.S.C. University Campus, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario